CLINICAL TRIAL: NCT00482599
Title: A Multicenter, Parallel Group, Comparative Trial Evaluating the Efficacy, Pharmacokinetics and Safety of Org 25969 in Subjects With Normal or Impaired Renal Function
Brief Title: Efficacy, Pharmacokinetics and Safety of Org 25969 in Subjects With Normal or Impaired Renal Function (19.4.304)(P05948)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05948; 19.4.304
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Anesthesia, General
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal renal function (Active Comparator): Org 25969 given to subjects with normal renal function
  Interventions: Drug: Sugammadex
- Impaired renal function (Experimental): Org 25969 given to subjects with impaired renal function
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Sugammadex — 2 mg/kg sugammadex administered intravenously at reappearance of T2 after 0.6 mg/kg rocuronium in patients with renal impairment and control patients
  Other Names: Org 25969

SUMMARY:
The purpose of this study is to compare the efficacy and pharmacokinetics of Org 25969 in subjects with normal or impaired renal function and to evaluate the safety of Org 25969 in subjects with impaired renal function.

ELIGIBILITY:
Inclusion Criteria:

* ASA class 1 - 3 for renally impaired patients, ASA class 1-2 for control group
* Age at least 18 years
* Scheduled for general anesthesia without further need for muscle relaxation other than one single dose of 0.6 mg.kg-1 rocuronium
* Scheduled for surgical procedures in the supine position
* Written informed consent
* Creatinine clearance (CLCR) < 30 mL/min for renally impaired group, CLCR = 80 mL/min for control group

Exclusion Criteria:

* Known or suspected neuromuscular disorders impairing NMB
* Known or suspected (family) history of malignant hyperthermia
* Known or suspected allergy to narcotics, muscle relaxants or other medication used during general anesthesia
* Use of medication known to interfere with NMBA based on the dose and the time of administration, such as antibiotics, anticonvulsants and Mg2+
* Pregnancy
* Childbearing potential without using any of the following methods of birth control: condom or diaphragm with spermicide, vasectomized partner ( > 6 months), intrauterine device, abstinence
* Breast-feeding
* Prior participation in any trial with Org 25969
* Participation in another clinical trial, not pre-approved by NV Organon, within 30 days of entering into trial 19.4.304, or for the UK only: Participation in another clinical trial, within 30 days of entering into trial 19.4.304.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-06-01 (Actual); Primary Completion 2006-04-13 (Actual); Study Completion 2006-04-13 (Actual)

PRIMARY OUTCOMES:
Time from start administration of Org 25969 to recovery T4/T1 ratio to 0.9 | After surgery

SECONDARY OUTCOMES:
Time from start administration of Org 25969 to recovery T4/T1 ratio to 0.7 and 0.8 | After surgery

REFERENCES:
- [Derived] Staals LM, Snoeck MM, Driessen JJ, van Hamersvelt HW, Flockton EA, van den Heuvel MW, Hunter JM. Reduced clearance of rocuronium and sugammadex in patients with severe to end-stage renal failure: a pharmacokinetic study. Br J Anaesth. 2010 Jan;104(1):31-9. doi: 10.1093/bja/aep340. PMID 20007792
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html